CLINICAL TRIAL: NCT00401895
Title: Clinical Efficacy of Transjugular Intrahepatic Portosystemic Shunt With 8- or 10-mm Covered Stents in Cirrhotic Patients: A Randomized Controlled Study
Brief Title: Transjugular Intrahepatic Portosystemic Shunt With 8- or 10-mm Covered Stents
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: An interim analysis revealed a significantly higher persistence/recurrence of complications of portal hypertension in the 8 mm-stent group.
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Riggio Oliviero, Department of Clinical Medicine Sapienza University of Rome
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ROMTIPSRCT
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Cirrhosis
Keywords: TRANSJUGULAR INTRAHEPATIC PORTOSYSTEMIC SHUNT; Covered stents; portal hypertension; hepatic encephalopathy
MeSH Terms: conditions — Fibrosis; Hypertension, Portal; Hepatic Encephalopathy

ARMS (2):
- 1 (Active Comparator): patients treated with 10 mm stent
  Interventions: Device: TIPS created with 8 or 10 mm covered stent
- 2 (Active Comparator): patients treated with 8 mm stent
  Interventions: Device: TIPS created with 8 or 10 mm covered stent

INTERVENTIONS:
Device: TIPS created with 8 or 10 mm covered stent — creation of a shunt between hepatic vein and portal vein with PTFE-covered stents
  Other Names: Viatorr Goretex

SUMMARY:
Coated stents with different diameters are presently commercially available, but clinical studies on the assessment of the best stent diameter for a better clinical efficacy, a reduced number of complications, and an effective portal pressure reduction (essential in the treatment of those pathologies in which TIPS is indicated) still do not exist.

Aim of the study The purpose of our study is to compare the clinical efficacy and the incidence of complications of TIPS created with 8- and 10-mm covered stents in patients with hepatic cirrhosis.

DETAILED DESCRIPTION:
Clinical Efficacy of Transjugular Intrahepatic Portosystemic Shunt With 8- or 10-mm Covered Stents in Cirrhotic Patients:

A Randomized Controlled Study

Introduction In the treatment of esophageal varices rebleeding1 and ascites/hydrothorax refractory to the diuretic therapy2 by transjugular intrahepatic portosystemic shunt (TIPS), shunt stenosis (occurring in 30-70% of cases during the first post-procedural year) and the onset of hepatic encephalopathy (30-55% of cases at one year) represent two major problems.

Since the year 2000, a new polytetrafluoroethylene covered stent has highly improved TIPS patency, thus inducing a remarkable reduction of rebleeding incidence. Some authors, however, suggest that the maintenance of the shunt patency may involve an increased risk of hepatic encephalopathy, although the data in the present literature are limited and controversial. The only randomized controlled study3 available, in fact, reports a lower incidence of hepatic encephalopathy in those patients treated with covered stents as compared with those treated with conventional metallic stents. In our preliminary experience,4 instead, a similar incidence of hepatic encephalopathy was noted in both groups. In addition, in the group of patients treated by covered stents, a higher number of cases with persistent and intractable hepatic encephalopathy (requiring shunt reduction) was recorded.5 Post-TIPS hepatic encephalopathy incidence increases with the decrease of post-procedure portal pressure which depends on the caliber of the stent used to create the anastomosis. This might suggest the use of covered stents with a smaller diameter aimed at reducing the risk of hepatic encephalopathy. Coated stents with different diameters are presently commercially available, but clinical studies on the assessment of the best stent diameter for a better clinical efficacy, a reduced number of complications, and an effective portal pressure reduction (essential in the treatment of those pathologies in which TIPS is indicated) still do not exist.

Aim of the study The purpose of our study is to compare the clinical efficacy and the incidence of complications of TIPS created with 8- and 10-mm covered stents in patients with hepatic cirrhosis.

Methods All consecutive cirrhotic patients who have undergone TIPS at our Department for bleeding of esophagogastric varices refractory to medical or endoscopic treatment or for ascites/hydrothorax refractory to diuretic therapy will be considered eligible for the study.

Before the TIPS procedure, all the patients will undergo a complete clinical evaluation (including psychometric tests) to assess their past or present history of hepatic encephalopathy; their Child-Pugh and MELD scores will be determined; abdominal ultrasounds and esophagogastroduodenoscopies will be also carried out. The patients will be then randomized into two groups to undergo TIPS with either 8- or 10-mm covered stents (VIATORR®, W. L. Gore & Associates Inc., Flagstaff, AZ). The two groups will be followed up according to the same post-TIPS protocol:

* an outpatient consultation one month post-procedure and every three months thereafter or when clinically necessary. Each consultation will include a clinical exam, Child-Pugh and MELD scores determination, and hepatic encephalopathy assessment;
* a post-procedure ultrasound will be carried out at one and four weeks, at three and six months, and every six months thereafter or in case of bleeding recurrence or ascites;
* a follow-up esophagogastroduodenoscopy will be performed at one week and at one month following TIPS, and every six months thereafter or when necessary;
* an angiography will be done in presence of shunt dysfunction (bleeding or ascites recurrence due portal hypertension) or in case of variceal recurrence at risk of bleeding associated with signs of shunt dysfunction at ultrasound.

The following study end-points are defined:

* hepatic encephalopathy incidence: the hepatic encephalopathy grade will be evaluated according to the modified West Haven Criteria. Those patients presenting grade II (lethargy, apathy, personality changes, inappropriate behavior, minimal disorientation for time or place) or higher grades of hepatic encephalopathy episodes will reach the main study end-point;
* incidence of persistent hepatic encephalopathy: defined as the presence of a continuous mental state alteration, with episodes of further worsening episodes;
* incidence of recurrent hepatic encephalopathy: defined as the onset of at least three episodes of open hepatic encephalopathy in a six-month period;
* incidence of variceal rebleeding: defined as the finding, at esophagogastroduodenoscopy, of ongoing or recent variceal hemorrhage or the finding of blood in the stomach and the presence of varices as the only potential cause of bleeding;
* shunt dysfunction: defined as the finding of a portosystemic gradient higher than 12 mm Hg and angiographic evidence of shunt stenosis or occlusion;
* recurrence of ascites: defined as the need of performing at least one evacuation of ascitic fluid with paracentesis;
* survival: all deaths of any cause will be recorded. All mortalities occurring within a six-week period from a digestive bleeding episode will be considered as related to the bleeding itself. All deaths occurring within 30 days post-TIPS placement will be considered as early mortality.

Sample size The sample size will be calculated on the main study end-point: the incidence of hepatic encephalopathy. On the basis of previous studies, the post-TIPS incidence of hepatic encephalopathy is considered to be of 50% at one year. To obtain a clinically significant (from 50 to 25%) encephalopathy incidence reduction (a = 5% and b= 20%) it will be therefore necessary to enroll 57 patients per group. Randomization will be by sealed envelopes in blocks of ten.

Statistical analysis The comparability of the two groups treated with 8- or 10-mm covered stents will be verified by c2 o Student t-test. The incidence of hepatic encephalopathy (main study end-point), shunt dysfunction, rebleeding, recurrence of ascites, and mortality (secondary end-points) will be calculated by Kaplan-Meier method and compared by Log-rank test. The Number Cruncher Statistical System (NCSS) software will be employed.

The rules and guidelines of the "Good Clinical Practice" and all legal requirements on sensitive data storage and experimental protocols will be followed.

References

1. Merli M, Salerno F, Riggio O, et al. Transjugular intrahepatic portosystemic shunt versus endoscopic sclerotheraphy for the prevention of variceal bleeding in cirrhosis: a randomized multicenter trial. Hepatology 1998; 27: 40-45.
2. Salerno F, Merli M, Riggio O, Cazzaniga M, Valeriano V, Pozzi M, Nicolini A, Salvatori F, and GIST. Randomized controlled study of TIPS versus paracentesis plus albumin in cirrhosis with severe ascites. Hepatology 2004; 40: 629-635.
3. Bureau C, Garcia-Pagan JC, Otal P, Pomier-Layrgrargues G, et al. Improved clinical outcome using polytetrafluoroethylene-coated stents for TIPS: results of a randomized study. Gastroenterology 2004; 126: 469-475.
4. Angeloni S, Merli M, Salvatori F, De Santis A, Fanelli F, Pepino D, Attili AF, Rossi P, Riggio O. Polytetrafluorethylene-covered stent-graft for TIPS procedure: 1-year patency and clinical results. Am J Gastroenterol 2004; 99:280-285.
5. Riggio O, Nicolao F, Angeloni S, Masini A, Salvatori F, Fanelli F, Efrati C, Merli M. Intractable hepatic encephalopathy after TIPS with polytetrafluoroethylene-covered stent-graft.

Scand J Gastroenterol 2003;38:570-2.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive cirrhotic patients who have undergone TIPS at our Department for bleeding of esophagogastric varices refractory to medical or endoscopic treatment or for ascites/hydrothorax refractory to diuretic therapy will be considered eligible for the study.

Exclusion Criteria:

* an age >75 years; past or present history of hepatic encephalopathy;
* a Z-score at trial making test-A (TMT-A) >1.5;
* bilirubine levels >5 mg/dl;
* creatinine levels >3 mg/dl;
* serious cardiac or pulmonary dysfunction;
* a Child-Pugh's score >11;
* a model end-stage liver disease (MELD) score >18;
* portal thrombosis;
* a diagnosis of hepatic carcinoma;
* sepsis;
* spontaneous bacterial peritonitis;
* renal insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
hepatic encephalopathy incidence: | 1 year

SECONDARY OUTCOMES:
incidence of persistent hepatic encephalopathy: defined as the presence of a continuous mental state alteration, with episodes of further worsening episodes; | one year
incidence of recurrent hepatic encephalopathy: defined as the onset of at least three episodes of open hepatic encephalopathy in a six-month period; | one year
incidence of variceal rebleeding: defined as the finding, at esophagogastroduodenoscopy, of ongoing or recent variceal hemorrhage or the finding of blood in the stomach and the presence of varices as the only potential cause of bleeding; | one year
shunt dysfunction: defined as the finding of a portosystemic gradient higher than 12 mm Hg and angiographic evidence of shunt stenosis or occlusion; | one year
recurrence of ascites: defined as the need of performing at least one evacuation of ascitic fluid with paracentesis; | one year
survival: all deaths of any cause will be recorded. All mortalities occurring within a six-week period from a digestive bleeding episode will be considered as related to the bleeding itself. All deaths occurring within 30 days post-TIPS placement will | one year

CONTACTS AND LOCATIONS:
Overall Officials: Oliviero Riggio, MD, Principal Investigator — Gastroenterology Unit
Locations (1):
- Gastroenterology Unit. dip. Medicina Clinica Policlinico Umberto I, Roma, Italy